CLINICAL TRIAL: NCT04689087
Title: A Prospective, Open-label, Single-arm Clinical Study Evaluating Tumor Treating Fields (TTFields) in Combination With Chemotherapy for Recurrent Glioblastom
Brief Title: A Prospective, Open-label, Single-arm Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yonggao Mou, Director of neurosurgery department, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: M-TTFields
Record Dates: First submitted 2020-12-08; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Recurrent Glioblastoma Multiforme
Keywords: recurrent GBM,; TTFields（Tumor Treating Fields）; chemotherapy
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Second line conventional treatment (Experimental)
  Interventions: Combination Product: TTFields

INTERVENTIONS:
Combination Product: TTFields — For patients with relapsed GBM, before receiving electric field treatment, the patient can be re-operated, and TTFields+BPC chemotherapy is used after surgery

SUMMARY:
the study is a prospective, single-arm, open-label trial, designed to explore the efficacy and safety of Tumor-Treating Fields (TTFields) combined with second-line chemotherapy treatment in recurrent glioblastoma multiforme (GBM) , TTFields is an portable, battery operated device for chronic treatment of patients with recurrent or progressive glioblastoma multiforme (GBM) using alternating electric fields

DETAILED DESCRIPTION:
PAST CLINICAL EXPERIENCE:

The effect of the electric fields generated by the TTFields has been tested in two Ⅲ phase trials in humans(EF-11&EF-14). The data from these trials suggest TTFields may improve time to disease progression and overall survival of recurrent GBM patients. EF-11 is a randomized, controlled trial, designed to test the efficacy and safety of a new medical device.Although the number of patients in the trials is small, FDA has approved TTFields as a therapy for patients with recurrent GBM.

DESCRIPTION OF THE TRIAL:

Patients with GBM whose disease has recurred or progressed despite standard treatment (Surgery, radiation therapy, Temozolomide treatment) and meet all of the requirements for participation in the study will be included.Before receiving TTFields treatment, the patient can receive surgery again, and TTFields+BPC chemotherapy can be used after surgery; TTFields+BPC chemotherapy can also be used directly without surgery.

During the trial, TTFields treatment is a cycle (treatment course) every four weeks, and patients are required to complete at least one cycle of treatment. Recommended average daily wearing time ≥18 hours, patients will need to return once every month the hospital outpatient clinics where they will be examined by a physician and undergo routine laboratory examinations. These routine visits will continue for as long as the patient's disease is not progressing. After progression, if such occurs, patients will need to return once per month for two more months to the outpatient clinic for similar follow up examinations.

During the visits to the clinic patients will be examined physically and neurologically. A routine MRI of the head will be performed at baseline and after 2, 4 and 6 months. After this follow up plan, patients will be contacted once per month by telephone to answer basic questions about their health status. If the disease progresses, imaging tumor assessment or survival follow-up will be performed every 2 months thereafter, until 12 months of follow-up.

The investigator will use the RANO evaluation criteria for tumor imaging assessment, and classify the objective tumor response as follows: The objective tumor response status based on the evaluation of the target lesion can be: complete response (CR), partial response (PR), stable disease ( SD), disease progression (PD).

SCIENTIFIC BACKGROUND:

Electric fields exert forces on electric charges similar to the way a magnet exerts forces on metallic particles within a magnetic field. These forces cause movement and rotation of electrically charged biological building blocks, much like the alignment of metallic particles seen along the lines of force radiating outwards from a magnet.

Electric fields can also cause muscles to twitch and if strong enough may heat tissues. TTFields are alternating electric fields of low intensity. This means that they change their direction repetitively many times a second. Since they change direction very rapidly (200 thousand times a second), they do not cause muscles to twitch, nor do they have any effects on other electrically activated tissues in the body (brain, nerves and heart). Since the intensities of TTFields in the body are very low, they do not cause heating.

The breakthrough finding made by NovoCure was that finely tuned alternating fields of very low intensity, now termed TTFields (Tumor Treating Fields), cause a significant slowing in the growth of cancer cells. Due to the unique geometric shape of cancer cells when they are multiplying, TTFields cause the building blocks of these cells to move and pile up in such a way that the cells physically explode. In addition, cancer cells also contain miniature building blocks which act as tiny motors in moving essential parts of the cells from place to place. TTFields cause these tiny motors to fall apart since they have a special type of electric charge.

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent prior to any procedure related to the study;
2. Recurrence and pathologically confirmed WHO Grade IV glioblastoma (GBM);
3. The tumor is located in the supratentorial area
4. Age ≥18 years;
5. Received radiotherapy and maintenance treatment with temozolomide;
6. Expected survival time: > 3 months;
7. KPS score ≥60;
8. Ability to comply with the plan;

Exclusion Criteria:

1. Other clinical trials are being tried
2. Had major surgery within 4 weeks before the start of the study or had not recovered after the surgery
3. Received radiotherapy within 4 weeks before the study
4. Received chemotherapy within 4 weeks before the study
5. Women during pregnancy;
6. Allergic to hydrogels;
7. There are important implants in the body, such as pacemaker, defibrillator, shunt tube, deep brain stimulator, etc.;
8. Patients with significantly increased intracranial pressure (shifted >5mm in imaging midline, obvious papilloma, nausea, vomiting, and decreased consciousness)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
OS6 | 6 months
  Overall survival at 6 months

SECONDARY OUTCOMES:
Overall survival at 12 months (OS12) | 12 months
  To evaluate the OS12 of patients with recurrent glioblastoma treated with TTFields combined with chemotherapy
overall survival OS(refers to the time from enrollment to tumor disease death from various causes) | 2 years
  To evaluate the OS of patients with recurrent glioblastoma treated with tumor electric field therapy combined with chemotherapy
Progression-free survival PFS | 2 years
  To evaluate the PFS of patients with recurrent glioblastoma treated with tumor electric field therapy combined with chemotherapy according to RANO standard
security | 2 years
  Adverse events and severe adverse events occurred during treatment were recorded by CTCAE V5.0, and the safety of tumor electric field therapy combined with chemotherapy was analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Yonggao Mu, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China